CLINICAL TRIAL: NCT03496025
Title: Mimetic Interfaces - Toispuoleisen Kasvohermohalvauksen Kojeellinen Kuntoutus Terveen Puolen Lihasaktiviteettiohjauksella. Stimulaattorin Prototyypin Testaus terveillä koehenkilöillä ja Kasvohermohalvauspotilailla.
Brief Title: Facial Function Reanimation by Electrical Pacing in Unilateral Facial Paralysis.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tampere University Hospital (Other)
Collaborators: Tampere University (Other); Tampere University of Technology (Other); Helsinki University Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R15067
Record Dates: First submitted 2018-03-19; First posted 2018-04-12 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2019-09

CONDITIONS: Facial Nerve Palsy
Keywords: facial nerve palsy; facial paralysis; functional electrical stimulation; facial pacing
MeSH Terms: conditions — Bell Palsy; Facial Paralysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electrical stimulation (Experimental)
  Interventions: Device: Electrical muscle stimulation

INTERVENTIONS:
Device: Electrical muscle stimulation — The intervention consists of activating paralyzed facial muscles with electrical stimulation.

SUMMARY:
Purpose of the trial is to study the activations of paralyzed facial muscles in a unilateral facial nerve palsy with a multi-channel electrical stimulator. The principle of the device is to measure muscle activity of the healthy side of the face by surface electromyography (EMG) and to use this information to stimulate the corresponding muscles of the paralyzed side. The ultimate goal is to develop a prosthetic device for persons with a facial nerve palsy.

The trial consists of several different studies. The studies' aims are 1. To study activations of paralyzed facial muscles by the electrical stimulation. 2. To study different stimulation pulse waveforms, frequencies, and electrode placement and their effect on the muscle activations and the tolerability of the stimulation. 3. To study whether a symmetrical movement on the paralyzed side can be achieved with electrical stimulation when compared to the movements of the healthy side. 4. To study tolerability of stimulation-elicited eye blink when watching a film and the effect of the stimulation-induced blink on the eye symptoms, the visual acuity, and the effects of the stimulation on the lacrimal fluid. 5. To develop a method for facial pacing, i.e. measuring the muscle activations on the healthy side of the face and to use this information to stimulate and activate the healthy side of the face.

Forty subjects with a chronic facial nerve palsy are recruited to the studies. Each subject can participate in one or several studies. Another forty subjects with an acute facial nerve palsy are recruited to the study on the tolerability and effect on the eye symptoms. Additionally, altogether ninety healthy volunteers are recruited to the studies in order to gather preliminary information on the tolerability and the effects of the stimulations.

ELIGIBILITY:
Inclusion Criteria:

* a unilateral peripheral facial nerve palsy (patients)
* willingness to participate (patients, healthy volunteers)

Exclusion Criteria:

* malignant diseases (a previously treated cancer is not an exclusion criterion)
* unstable cardiovascular disease
* severe immune deficiency
* other severe neurological diseases (causing cognitive or physical impairment)
* diabetic neuropathy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Amplitudee of the movement elicited by electrical stimulation | Immediate
  The offline video analysis is done to determine the current threshold at which a movement of the target muscle is produced. Possible activations of the other muscles alongside the target muscle are also observed. The amplitude of the movement is analyzed offline from a video recording either visually by the investigators, or measured with a digital ruler. With visual evaluation, the outcome is measured on a rough level, i.e. whether the stimulated movement was larger in amplitude compared to the voluntary movement. With a digital ruler, the results a presented numerically (millimeters). The stimulated activation is compared to the voluntary activation of the muscle. Further, in some sub-studies, the facial activations are evaluated with the Facial Action Coding System.

SECONDARY OUTCOMES:
Subjective ratings related to the tolerability of stimulations | Immediate
  The participants evaluate the experienced discomfort and painfulness of the stimulation with a numeric rating scale (NRS).
Subjective ratings related to acceptability of the stimulated movement | Immediate
  The participants evaluate the naturalness and symmetry and their satisfaction with the stimulation elicited movement with an NRS.
Visual acuity | Immediate
  In substudies concerning the elicitation of eye blink, The visual acuity is measured for both eyes separately with a LogMAR chart before and after the stimulation session.
Changes in lacrimal fluid | Immediate
  In substudies concerning the elicitation of eye blink, a lacrimal fluid sample is collected before and after the stimulation session to investigate the possible effects of the stimulation in its constitution.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Rautiainen, MD, PhD, Study Director — professor, head physician
Locations (1):
- Tampere University Hospital, Tampere, Finland

REFERENCES:
- [Derived] Makela EA, Ilves MK, Venesvirta HM, Lylykangas JK, Rantanen VT, Vehkaoja AT, Verho JA, Lekkala J, Surakka VV, Rautiainen MEP. Effect of pulse waveforms on movement amplitudes and perceived discomfort in electric muscle stimulation in unresolved facial nerve palsy. Biomed Phys Eng Express. 2020 Mar 25;6(3):035013. doi: 10.1088/2057-1976/ab7eea. PMID 33438658